CLINICAL TRIAL: NCT06707935
Title: Is a Picture Worth a Thousand Words: A Participatory Approach to Codesign Descriptive and Pictorial Social Norm Nudges and a Randomised Controlled Trial (RCT) to Examine Their Effectiveness in Improving Mental Health Help-seeking Intention
Brief Title: Mental Health Help-seeking Promotion in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, LIU Tianyin Bridget, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSEARS20231109001
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Mental Health Help-seeking
Keywords: co-design; nudge; behavioural economics; mental health; help-seeking
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Descriptive social norm nudges (Experimental): Participants receive messages with social norm nudges presented in the word form.
  Interventions: Behavioral: Descriptive social norm nudges
- Pictorial social norm nudges (Experimental): Participants receive messages with social norm nudges presented in graphic form.
  Interventions: Behavioral: Pictorial social norm nudges
- Active control (Active Comparator): Participants receive messages with generic mental health knowledge or information.
  Interventions: Behavioral: Service as usual

INTERVENTIONS:
Behavioral: Descriptive social norm nudges — A set of messages with descriptive social norm nudges sent to participants.
  Arms: Descriptive social norm nudges
Behavioral: Pictorial social norm nudges — A set of messages with pictorial social norm nudges sent to participants.
  Arms: Pictorial social norm nudges
Behavioral: Service as usual — Traditional mental health education information disseminated to participants.
  Arms: Active control

SUMMARY:
The present study aims to examine the effectiveness of descriptive social norm nudges and pictorial social norm nudges in improving mental health help-seeking intention compared to educational information.

DETAILED DESCRIPTION:
This study is a three-arm randomised controlled trial (RCT) in 540 older adults aged 60 years and above recruited through NGOs, testing the utility of revised TPB with baseline data, and the effectiveness of descriptive social norm-nudges (intervention group 1) and pictorial social norm- nudges (intervention group 2) comparing to traditional mental health education (control). Participants will be evenly randomised and receive 1 message/picture per day consecutively for 2 weeks. Researchers blind to group allocation will interview participants at baseline (T0), 2 weeks (post-intervention, T1), and 12 weeks (follow-up, T2). The primary outcomes are changes in subjective norms and help-seeking intention assessed using a revised Chinese version of the theory of planned behaviour questionnaire (C-TPB); secondary outcomes include perceived behavioural control, help-seeking attitude, perceived barriers to help-seeking (C-TPB subscales), and mental health assessed by PHQ-9, GAD-7 and UCLA-3.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 years or above at the time of the baseline assessment
* have no severe mental disorder or cognitive impairment
* have no severe visual impairment
* be able to read Chinese
* have a smartphone with an instant communication application to receive text and images

Exclusion Criteria:

* have severe difficulty in reading and communication
* show imminent suicidal risk at any stage of the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Subjective norms toward mental health help-seeking | Baseline (T0), post-intervention (T1, two weeks after T0), and to 12 weeks after the baseline (T2)
  Subjective norms toward mental health help-seeking will be measured by six items adapted from the validated Chinese version of the TPB questionnaire (C-TPB) . The three items will measure descriptive norms describing what society, in general, does when facing mental health challenges, and the other three items will measure social norms describing what the significant others of the participant would do. Responses will be rated on a 6-point Likert scale, with higher scores indicating higher levels of subjective norms about mental health help-seeking.
Mental health help-seeking intention | Baseline (T0), post-intervention (T1, two weeks after T0), and to 12 weeks after the baseline (T2)
  Mental health help-seeking intention will be measured on a 3-item subscale of C-TPB. Responses will be rated on a 6-point Likert scale, with higher scores indicating higher levels of help-seeking intention.

SECONDARY OUTCOMES:
Perceived behavioural control | Baseline (T0), post-intervention (T1, two weeks after T0), and to 12 weeks after the baseline (T2)
  Perceived behavioural control will be measured on a 3-item subscale of the C-TPB. Responses are rated on a 6-point Likert scale, with higher scores indicating higher levels of behavioural control.
Help-seeking attitude | Baseline (T0), post-intervention (T1, two weeks after T0), and to 12 weeks after the baseline (T2)
  Help-seeking attitude will be measured on a 5-item subscale of C-TPB, items will be measured on a 6-point semantic differential scale, with higher scores indicating a more positive attitude towards help-seeking.
Perceived barriers to help-seeking | Baseline (T0), post-intervention (T1, two weeks after T0), and to 12 weeks after the baseline (T2)
  Perceived barriers to help-seeking will be measured by a 6-item scale adapted from the Chinese American Psychiatric Epidemiological study (CAPES), responses are rated on a 6-point Likert scale, with higher scores indicating more significant perceived barriers to help-seeking.
Depressive symptoms | Baseline (T0), post-intervention (T1, two weeks after T0), and to 12 weeks after the baseline (T2)
  Depressive symptoms will be measured with the Patient Health Questionnaire (PHQ-9). It is a 9-item instrument that incorporates depression diagnostic criteria with other leading major depressive symptoms and rates the frequency of the symptoms, factoring into the scoring severity index. PHQ-9 scores of 5-9, 10-14, 15-19, 20 and above represent mild, moderate, moderately severe, and severe depression, respectively.
Anxiety symptoms | Baseline (T0), post-intervention (T1, two weeks after T0), and to 12 weeks after the baseline (T2)
  Anxiety will be measured with the Generalised Anxiety Disorder 7-item scale (GAD-7). It is a 7-item scale; responses to each item are rated on a 4-point Likert scale and range from 0 to 3. It taps on the most prominent diagnostic features for GAD, and scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate, and severe anxiety, respectively.
Loneliness | Baseline (T0), post-intervention (T1, two weeks after T0), and to 12 weeks after the baseline (T2)
  Loneliness will be measured with the UCLA Loneliness Scale (UCLA-3). It is a 3-item scale measuring an individual's perceived loneliness. Each item is evaluated with scores ranging from 0 (never) to 3 (often), the total score is the sum of all items, and a higher score indicates a higher level of perceived loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Tianyin Liu, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT06707935/Prot_SAP_000.pdf